CLINICAL TRIAL: NCT02805907
Title: Efficacy of Calcifediol Supplementation in Asthma Control in Asthmatic Patients With Vitamin D Deficiency (ACViD)
Acronym: ACViD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MurciaSalud (Other Government)
Responsible Party: Principal Investigator, Rubén Andújar, Medical Doctor. Pulmonologist, MurciaSalud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 300681
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-04

CONDITIONS: Asthma, Bronchial
MeSH Terms: conditions — Asthma | interventions — Calcifediol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (IG) (Experimental): Calcifediol (Hidroferol®) in 16,000-IU ampoules taken weekly by the oral route
  Interventions: Drug: Calcifediol
- Control Group (CG) (Placebo Comparator): Placebo in a presentation with an identical appearance taken weekly by the oral route
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcifediol
  Arms: Intervention Group (IG)
Drug: Placebo
  Arms: Control Group (CG)

SUMMARY:
Introduction: There are many cross-sectional studies in children and adults indicating that low vitamin D levels in asthmatic patients are correlated with poorer asthma control, poorer lung function, decreased response to glucocorticoids and more frequent exacerbations. Moreover, as there is a significant group of asthmatic patients having insufficient control of their disease, despite high doses of inhaled corticosteroids, we have investigated new treatment alternatives, which include vitamin

Objective: To determine the efficacy of vitamin D supplementation in asthmatic patients with vitamin D deficiency in degree of asthma control.

Materials and methods: A prospective, controlled, randomised, triple-blind study was conducted with a follow-up of 6 months. The patients recruited were over 18 years of age with a medical diagnosis of bronchial asthma and serum 25(OH)D3 levels < 30 ng/ml. Patients were excluded if they had a smoking habit ≥ 10 pack-years, taking vitamin D supplements, kidney disease (creat. > 2 mg/dl), hypercalcaemia (corrected with proteins > 10.5 mg/dl), a repeat episodes of renal colic, any gastrointestinal disease that might interfere with vitamin D absorption, or severe psychosocial problems, or were pregnant or breast-feeding. The randomisation process assigned patients to one of two groups: a group that received vitamin D (in the form of calcifediol (Hidroferol®) in 16,000-IU ampoules taken weekly by the oral route) and another group that received placebo in a presentation with an identical appearance and the same administration regimen. Demographic, clinical, spirometry and laboratory endpoints were collected. The primary endpoint was degree of asthma control as determined by the internationally validated Asthma Control Test (ACT). The secondary endpoints were asthma exacerbations, dose of inhaled corticosteroids and quality of life as measured using the Mini-AQLQ (Asthma Quality of Life Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of bronchial asthma
* serum 25(OH)D3 levels < 30 ng/ml.

Exclusion Criteria:

* smoking habit ≥ 10 pack-years,
* taking vitamin D supplements,
* kidney disease (creat. > 2 mg/dl),
* hypercalcaemia (corrected with proteins > 10.5 mg/dl),
* repeat episodes of renal colic,
* any gastrointestinal disease that might interfere with vitamin D absorption,
* severe psychosocial problems,
* pregnant
* breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Andújar Espinosa, Medicine, Principal Investigator — MurciaSalud
Locations (1):
- Servicio Murciano de Salud, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castro M, King TS, Kunselman SJ, Cabana MD, Denlinger L, Holguin F, Kazani SD, Moore WC, Moy J, Sorkness CA, Avila P, Bacharier LB, Bleecker E, Boushey HA, Chmiel J, Fitzpatrick AM, Gentile D, Hundal M, Israel E, Kraft M, Krishnan JA, LaForce C, Lazarus SC, Lemanske R, Lugogo N, Martin RJ, Mauger DT, Naureckas E, Peters SP, Phipatanakul W, Que LG, Sheshadri A, Smith L, Solway J, Sullivan-Vedder L, Sumino K, Wechsler ME, Wenzel S, White SR, Sutherland ER; National Heart, Lung, and Blood Institute's AsthmaNet. Effect of vitamin D3 on asthma treatment failures in adults with symptomatic asthma and lower vitamin D levels: the VIDA randomized clinical trial. JAMA. 2014 May;311(20):2083-91. doi: 10.1001/jama.2014.5052. PMID 24838406
- [Derived] Andujar-Espinosa R, Salinero-Gonzalez L, Illan-Gomez F, Castilla-Martinez M, Hu-Yang C, Ruiz-Lopez FJ. Effect of vitamin D supplementation on asthma control in patients with vitamin D deficiency: the ACVID randomised clinical trial. Thorax. 2021 Feb;76(2):126-133. doi: 10.1136/thoraxjnl-2019-213936. Epub 2020 Nov 5. PMID 33154023

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group (IG): Calcifediol (Hidroferol®) in 16,000-IU ampoules taken weekly by the oral route
  Calcifediol
- Control Group (CG): Placebo in a presentation with an identical appearance taken weekly by the oral route
  Placebo
Period: Overall Study
Arm/Group | Intervention Group (IG) | Control Group (CG)
Started | 56 | 56
Completed | 53 | 53
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (IG) | Control Group (CG) | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.57 (15.83) | 56.61 (15.00) | 55.59 (15.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 47 | 87
  Male | 16 | 9 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 56 | 56 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 56 | 56 | 112
Initial Asthma Control Test (ACT) [Mean (Standard Deviation); unit: units on a scale] — Interpretation of the ACT questionnaire: Score less than or equal to 15 points: poor control; Between 16 and 19 points: partially controlled; Greater or equal to 20 points: good control.
  units on a scale | 17.71 (4.54) | 19.02 (4.59) | 18.37 (4.59)
Initial Asthma Quality of Life Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The response options for each item are placed on an equidistant 7-point scale, where 1 = maximum limitation and 7 = no limitation. The questionnaire Global score, which is the mean for all 15 items that make up the scale, and a score for each dimension, which is the average of the corresponding items for that dimension.
  units on a scale | 4.38 (1.62) | 4.85 (1.96) | 4.62 (1.91)
Asthma Severity [Count of Participants; unit: Participants]
  Intermitent | 5 | 12 | 17
  Mild Persistent | 9 | 11 | 20
  Moderate Persistent | 29 | 27 | 56
  Severe Persistent | 13 | 6 | 19
Exacerbations [Mean (Standard Deviation); unit: Exacerbations in the last 6 months] — Number of exacerbations in the last 6 months
  Exacerbations in the last 6 months | 1.18 (1.55) | 1.14 (2.70) | 1.16 (2.19)
Hospitalizations [Mean (Standard Deviation); unit: Hospitalizations in the last 6 months] — Number of hospitalizations in the last 6 months
  Hospitalizations in the last 6 months | 0.11 (0.31) | 0.13 (0.33) | 0.12 (0.32)
Emergency care [Mean (Standard Deviation); unit: Emergency care in the last 6 months] — Number of emergency care in the last 6 months
  Emergency care in the last 6 months | 0.45 (0.81) | 0.59 (1.30) | 0.52 (1.08)

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Measured With Asthma Control Test (ACT)
Description: Asthma Control Test (ACT): Interpretation of the ACT questionnaire: Score less than or equal to 15 points: poor control; Between 16 and 19 points: partially controlled; Greater or equal to 20 points: good control.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group (IG) | Control Group (CG)
Number analyzed (Participants) | 53 | 53
units on a scale | 20.49 (4.13) | 18.23 (5.70)

2. Secondary Outcome: Number of Asthma Exacerbations
Description: Number of asthma exacerbations during the study period
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Asthma exacerbations
Arm/Group | Intervention Group (IG) | Control Group (CG)
Number analyzed (Participants) | 53 | 53
Asthma exacerbations | 1 (0.20) | 0 (0.4)

3. Secondary Outcome: Dose Inhaled Corticosteroids as the Scale of the Spanish Guide for Asthma Management (GEMA 4.0)
Description: Dose inhaled corticosteroids as the scale of the Spanish guide for asthma management (GEMA 4.0): Depends on the type of steroids:
  Beclomethasone dipropionate (Low dose: 200-500 mcg/day, Half dose: 501-1000 mcg/day, High dose: 1001-2000 mcg/day), Beclomethasone extrafine (Low dose: 100-200 mcg/day, Half dose: 201-400 mcg/day, High dose: > 400 mcg/day), Budesonide (Low dose: 200-400 mcg/day, Half dose: 401-800 mcg/day, High dose: 801-1600 mcg/day), Ciclesonide (Low dose: 80-160 mcg/day, Half dose: 161-320 mcg/day, High dose: 321-1280 mcg/day), Fluticasone furoate (Half dose: 92 mcg/day, High dose: 184 mcg/day), Fluticasone propionate (Low dose: 100-250 mcg/day, Half dose: 251-500 mcg/day, High dose: 501-1000 mcg/day), Mometasone furoate (Low dose: 100-200 mcg/day, Half dose: 201-400 mcg/day, High dose: 401-800 mcg/day),
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (IG) | Control Group (CG)
Number analyzed (Participants) | 53 | 53
Participants
  Low | 18 | 24
  Half | 30 | 23
  High | 5 | 6

4. Secondary Outcome: Quality of Life Measured With Mini-AQLQ (Asthma Quality of Life Questionnaire)
Description: Mini-AQLQ (Asthma Quality of Life Questionnaire): The response options for each item are placed on an equidistant 7-point scale, where 1 = maximum limitation and 7 = no limitation. The questionnaire Global score, which is the mean for all 15 items that make up the scale, and a score for each dimension, which is the average of the corresponding items for that dimension.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group (IG) | Control Group (CG)
Number analyzed (Participants) | 53 | 53
units on a scale | 5.34 (1.29) | 4.64 (1.56)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention Group (IG) | Control Group (CG)
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 3/56 | 2/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (IG) (N=56) | Control Group (CG) (N=56)
dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No